CLINICAL TRIAL: NCT00639470
Title: Parents Reading Comprehension of Their Child's Post-Operative Medicine Fact
Brief Title: Parents Reading Comprehension of Their Child's Post-Operative Medicine Fact Sheets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sharon Kitchie, PhD, APRN, BC, SUNY Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRBPHS#5229
Record Dates: First submitted 2008-03-12; First posted 2008-03-20 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Parents
Keywords: Patient Education Handout; Parents; Patient Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: easy to read fact sheets — easy to read fact sheets with illustrations and without illustrations
  Other Names: patient education handouts

SUMMARY:
The objective of this study is to test legal guardians reading comprehension of their child's post-operative medication administration using three different versions of written medication information (standard fact sheets, easy-to-read fact sheets, and easy-to-read fact sheets accompanied by illustrations).

DETAILED DESCRIPTION:
It is important for the child's welfare and comfort that the legal guardian can read and comprehend their child's pain medication information. Failure to understand the full implications of the medication may jeopardize the child's comfort level or welfare. Readability of printed education materials is a key to comprehension and supplements what healthcare providers verbally tell the parents/legal guardians. Several studies have demonstrated the benefits of using illustrations to convey intended messages. Simple line drawings appear to do well with those who have low-literacy skills.

The following hypothesis will be tested:

* There is no difference in level of comprehension of medication administration by the legal guardians who receive standard fact sheets about medication, those who receive easy-to-read fact sheets, and those who receive easy-to-read fact sheets accompanied by illustrations.
* There is no difference in level of comprehension of pain assessment by the legal guardians who receive standard fact sheets about assessing pain, those who receive easy-to-read fact sheets, and those who receive easy-to-read facts sheets accompanied by illustrations.
* There is no relationship between legal guardians' satisfaction with medication education and whether they receive standard fact sheets, easy-to-read fact sheets, or those who receive easy-to read fact sheets accompanied by illustrations.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years of age or older or an emancipated minor
* ability to see, speak, and hear English
* have a child who will be undergoing surgery
* signed surgical consent form
* have a child staying on hospital pediatric surgical unit after surgery until discharge
* have a child admitted for at least one day but not more than 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-08; Primary Completion 2007-03 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Comprehension of the fact sheets as measured by the Cloze Readability Procedure. | On the day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Kitchie, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States